CLINICAL TRIAL: NCT02013128
Title: A Multi-center Phase II Study With Safety Run-in Evaluating the Efficacy and Safety of Ublituximab in Combination With Ibrutinib in Patients With Select B-Cell Malignancies
Brief Title: Ublituximab + Ibrutinib in Select B-cell Malignancies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: TG Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UTX-IB-104
Record Dates: First submitted 2013-12-11; First posted 2013-12-17 (Estimated); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Chronic Lymphocytic Leukemia; Mantle Cell Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Mantle-Cell | interventions — ublituximab; ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ublituximab + ibrutinib (Experimental): Ublituximab: IV infusion dose Days 1, 8 and 15 followed by maintenance infusions Ibrutinib: Fixed oral daily dose
  Interventions: Drug: Ublituximab; Drug: Ibrutinib

INTERVENTIONS:
Drug: Ublituximab — Ublituximab (IV infusion)
Drug: Ibrutinib — Ibrutinib oral daily dose
  Other Names: Ibrutinib (IMBRUVICA)

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of Ublituximab in combination with Ibrutinib in patients with advanced hematologic malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed Mantle Cell lymphoma (MCL) open for enrollment. The Chronic Lymphocytic Leukemia (CLL) enrollment arm is now closed.
* Refractory to or relapsed after at least 1 prior treatment regimen
* Eastern Cooperative Oncology Group (ECOG) score of 0 to 2

Exclusion Criteria:

* Any major surgery, chemotherapy or immunotherapy within the last 21 days
* Known hepatitis B virus, hepatitis C virus or HIV infection
* Autologous hematologic stem cell transplant within 3 months of study entry. Prior Allogeneic hematologic stem cell transplant is excluded.
* Richter's transformation, prolymphocytic leukemia or primary central nervous system lymphoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2014-01-06 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of ublituximab in combination with ibrutinib in patients with select B-cell malignancies | 28 days (1 cycle of therapy)
  To determine the incidence of adverse events, any potential abnormal laboratory results and any dose-limiting toxicities

SECONDARY OUTCOMES:
Overall Response Rate | Up to 1 year
  To assess the overall response rate (ORR) in patients with hematologic malignancies treated with Ublituximab in combination with Ibrutinib

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Sharman, MD, Study Chair — Willamette Valley Cancer Institute
Locations (18):
- United States (18):
  - TG Therapeutics Investigational Trial Site, Huntsville, Alabama
  - TG Therapeutics Investigational Trial Site, Tucson, Arizona
  - TG Therapeutics Investigational Trial Site, Santa Barbara, California
  - TG Therapeutics Investigational Trial Site, Boulder, Colorado
  - TG Therapeutics Investigational Trial Site, Niles, Illinois
  - TG Therapeutics Investigational Trial Site, Urbana, Illinois
  - TG Therapeutics Investigational Trial Site, Bethesda, Maryland
  - TG Therapeutics Investigational Trial Site, Morristown, New Jersey
  - TG Therapeutics Investigational Trial Site, Portland, Oregon
  - TG Therapeutics Investigational Trial Site, Springfield, Oregon
  - TG Therapeutics Investigational Trial Site, Greenville, South Carolina
  - TG Therapeutics Investigational Trial Site, Memphis, Tennessee
  - TG Therapeutics Investigational Trial Site, Austin, Texas
  - TG Therapeutics Investigational Trial Site, Dallas, Texas
  - TG Therapeutics Investigational Trial Site, Tyler, Texas
  - TG Therapeutics Investigational Trial Site, Blacksburg, Virginia
  - TG Therapeutics Investigational Trial Site, Fairfax, Virginia
  - TG Therapeutics Investigational Trial Site, Vancouver, Washington